CLINICAL TRIAL: NCT03068182
Title: Cardiovascular Responses to Arm Crank Exercise Versus to Treadmill Exercise in Adult Subjects
Brief Title: Effects of Arm Crank Versus Treadmill Exercises on Heart Rate Variability in Adult Subjects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Alsayed Abd Elhameed Shanb, Associate professor, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2015-03-159
Record Dates: First submitted 2017-02-26; First posted 2017-03-01 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-02

CONDITIONS: Heart Rate Variability
Keywords: Exercise ,Autonomic cardiac function ,Adult subjects
MeSH Terms: interventions — Exercise Test; Exercise

STUDY DESIGN:
Intervention Model Description: Parallel assignments
Who Masked: Participant, Investigator
Masking Description: by a blinded and independent research assistant who opened sealed envelopes that contained a computer-generated randomization card
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm crank Exercise (Experimental): Sixty-five participated in an arm crank moderate intensity exercise for 40 minutes.
  Interventions: Device: Arm crank; Other: Exercise
- Treadmill Exercise (Experimental): Sixty-five participated in a treadmill moderate intensity exercise for 40 minutes.
  Interventions: Device: Treadmill; Other: Exercise

INTERVENTIONS:
Device: Arm crank — Each participant practiced on arm crank (Hudson) from long sitting position for 40 minutes. Seat's height and distance were adjusted to achieve full extension of subject arms at horizontal shoulder-level position
  Arms: Arm crank Exercise
Device: Treadmill — Participant practiced on an electronic computerized treadmill for 40 minutes . participant began warming up with lowest speed treadmill exercise for 5 minutes at zero inclination. Treadmill speed was increased gradually to achieve the pre-determined individualized moderate intensity for 30 minutes
  Arms: Treadmill Exercise
Other: Exercise

SUMMARY:
Cardiovascular response to exercise affects the capacity of all body organs depending upon intensity, duration and mode of exercises. The aim was to compare acute effects of arm crank with treadmill moderate intensity exercises on heart rate variability in normal participants.

DETAILED DESCRIPTION:
A one hundred thirty male volunteers were equally and randomly assigned to; Group-I: Sixty-five participated in an arm crank moderate intensity exercise for 40 minutes. Group-II: Sixty-five participated in a treadmill moderate intensity exercise for 40 minutes. Halter heart rate monitor and automatic sphygmomanometer were used to measure heart beat intervals and arterial blood pressure respectively.

ELIGIBILITY:
Inclusion Criteria:

* Normal adult non-obese male subjects , their age ranges from 25-36 years.
* They were asymptomatic for cardiovascular and respiratory diseases.
* They currently did not receive any medical prescriptions.
* All participants were asked to avoid strenuous exercise, give up caffeine and alcohol beverages to have sufficient rest for 2 days before measurement sessions to avoid any carry over effects of stimulants or depressants on autonomic functions

Exclusion Criteria:

* Any participant had medical history of cardiovascular and pulmonary disorders or received any interfering medications with study was excluded

Ages: 25 Years to 36 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-09-25 (Actual); Study Completion 2017-01-25 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | 45 minutes
  Autonomic functions of the heart was measured

SECONDARY OUTCOMES:
Blood pressure | 5 minutes
  Arm blood pressure was measured

CONTACTS AND LOCATIONS:
Overall Officials: Alsayed A Shanb, PhD, Principal Investigator — Imam Abdulrahman Bin Faisal University; Enas F Youssef, PhD, Study Director — Imam Abdulrahman Bin Faisal University
Locations (1):
- University of Dammam, Dammam, Estern Pronince, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
The final comment of our results only will be shared

REFERENCES:
- [Result] White DW, Raven PB. Autonomic neural control of heart rate during dynamic exercise: revisited. J Physiol. 2014 Jun 15;592(12):2491-500. doi: 10.1113/jphysiol.2014.271858. Epub 2014 Apr 22. PMID 24756637
- See also: Description it is a scientific location — https://jyx.jyu.fi/dspace/handle/123456789/37910